CLINICAL TRIAL: NCT00241657
Title: Immune Responses to BCG Vaccination in Malawi and the UK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KPS10
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2002-12

CONDITIONS: Immunity, Cellular; Hypersensitivity, Delayed Type
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: BCG

SUMMARY:
BCG vaccination has been found to provide greater protection against TB in the UK than in Malawi. This study compares immune responses in BCG-vaccinated and unvaccinated teenagers and young adults in Malawi and in the UK.

ELIGIBILITY:
Inclusion Criteria:

* BCG unvaccinated
* HIV negative
* Not pregnant
* Informed Consent

Exclusion Criteria:

* HIV positive
* Pregnant
* Seriously ill

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

PRIMARY OUTCOMES:
Delayed-type hypersensitivity
cytokine responses (eg IFNg) to mycobacterial antigens

SECONDARY OUTCOMES:
scar size

CONTACTS AND LOCATIONS:
Overall Officials: Paul EM Fine, VMD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Karonga Prevention Study, Chilumba, Karonga District, Malawi
- Redbridge and Waltham Forest Primary Care Trust, Ilford, Essex, United Kingdom